CLINICAL TRIAL: NCT00184145
Title: EMDR (Eye Movement Desensitization and Reprocessing) in the Treatment of Specific Phobia. A Randomised Controlled Trial.
Brief Title: EMDR in the Treatment of Specific Phobia.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: approval of ethical committee was denied
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPLK-2004
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Specific Phobia
Keywords: Specific (Animal) Phobia; EMDR; Exposure therapy
MeSH Terms: conditions — Phobia, Specific; Phobic Disorders | interventions — Eye Movement Desensitization Reprocessing; Implosive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EMDR (Experimental): The experimental group was treated for animal phobia by EMDR, control group received an attention placebo (relaxation plus breathing exercises). Afterwards, both groups were treated by exposure therapy (therapy of choice for animal phobia).
  Interventions: Other: EMDR (Eye Movement Desensitization and Reprocessing); Other: Exposure therapy

INTERVENTIONS:
Other: EMDR (Eye Movement Desensitization and Reprocessing) — Psychotherapy which is approved for PTSD.
Other: Exposure therapy — All participants in the study received exposure therapy som second treatment. Exposure therapy is the therapy of choice for animal phobia.

SUMMARY:
The purpose for this study is to determine whether EMDR is effective in the treatment of specific (animal) phobia.

DETAILED DESCRIPTION:
Aims: To test the hypothesis that one session EMDR is more effective for the treatment of specific (animal) phobia than relaxation immediately after treatment and at follow-up. Secondly to test whether an additional one-session exposure therapy offered to both treatment groups (EMDR patients and relaxation patients) improves outcome in the EMDR-group and results in equal outcome for both treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Specific (Animal) Phobia

Exclusion Criteria:

* Current or past psychotic disorder
* Current substance dependence or abuse
* Serious physical illness
* Active suicidal behavior
* Bipolar affective disorder
* Pregnancy

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-06 (Actual); Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Behavioral Approach Test towards the feared animal. | Before and after each treatment

SECONDARY OUTCOMES:
Scores on self-report questionnaires on phobic symptoms | Before and after both treatments
Neuropsychological function | Before first treatment, some measures also before second treatment
Cognitive strategies | Before both treatments

CONTACTS AND LOCATIONS:
Overall Officials: Ludger Kaiser, Doctor, Principal Investigator